CLINICAL TRIAL: NCT00732888
Title: Effect of Calcium Supplements on Nilotinib Hydrochloride Pharmacokinetics in Healthy Volunteers (CAMN107DUS10T) (UPCI 08-077)
Brief Title: Effect of Calcium on Tasigna Pharmacokinetics (PK) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jan Beumer (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Jan Beumer, Principal Investigator, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 08-077; CAMN107DUS10T; UPCI 08-077
Record Dates: First submitted 2008-08-07; First posted 2008-08-12 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Healthy
Keywords: Pharmacokinetics; Healthy volunteers; No condition; Pharmacokinetics study
MeSH Terms: interventions — nilotinib; Calcium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): On an 18-day schedule, calcium supplement (Tums Ultra 1000®) once daily on day 15; and Tasigna® once daily on days 1 and 15 (i.e., Tasigna® alone on day 1, and combination of Tasigna® and calcium supplement on day 15).
  Interventions: Drug: Nilotinib Hydrochloride; Dietary Supplement: calcium carbonate
- 2 (Other): On an 18-day schedule, calcium supplement (Tums Ultra 1000®) once daily on day 1; and Tasigna® once daily on days 1 and 15 (i.e., combination of Tasigna® and calcium supplement on day 1, Tasigna® alone on day 15).
  Interventions: Drug: Nilotinib Hydrochloride; Dietary Supplement: calcium carbonate

INTERVENTIONS:
Drug: Nilotinib Hydrochloride — Dosage form: capsules Dosage: 400 mg (2 x 200 mg capsule) Frequency & duration: On an 18-day schedule, one dose administered once on day 1 and once on day 15 (2 doses total)
  Other Names: Tasigna®; AMN107
Dietary Supplement: calcium carbonate — Dosage form: tablets Dosage: 4000 mg (4 x 1000 mg tablet) Frequency: On an 18-day schedule, once daily day 15 (for Arm 1); or once daily day 1 (for Arm 2)
  Other Names: Tums Ultra 1000®

SUMMARY:
This research study is being conducted through the University of Pittsburgh Cancer Institute (UPCI). It will evaluate the concentrations of Tasigna®, an oral drug used to treat some types of cancer, in the blood of healthy volunteers when taken with and without Tums Ultra®, a calcium product often used in the treatment of upset stomach and as a calcium supplement.

DETAILED DESCRIPTION:
This is an open-label, single-institution, randomized cross-over, fixed-schedule investigation of the effects of calcium carbonate on the pharmacokinetics (PK) of Tasigna® in healthy volunteers. Healthy volunteers will be recruited to participate in this study such that twelve subjects (6 men / 6 women) will complete the study at UPCI. Subjects will be compensated for participation.

Half of the subjects will receive Tasigna® alone on Day 1 and Tasigna® and calcium carbonate on Day 15, and the other half will receive Tasigna® and calcium carbonate on Day 1 and Tasigna® alone on Day 15, determined by randomization of subjects receiving either the combination or Tasigna® alone during the first visit. Doses will be 400 mg Tasigna® (2 x 200 mg tablets) and 4000 mg calcium carbonate (4 x Tums Ultra 1000® chewable tablets, equivalent to 4000 mg calcium carbonate or 1600 mg calcium).

Multiple PK blood samples will be taken from Days 1-4 and Days 15-18. Tasigna® PK will be assessed after oral administration of 400 mg Tasigna® alone, and after oral administration of 400 mg Tasigna® with concomitant administration of 4000 mg calcium carbonate. Two two-day/one-night inpatient stays and four brief outpatient visits are required to accommodate all study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women 18 years of age or older. Healthy subjects are defined as individuals who are free from clinically significant illness or disease (such as coronary arterial disease, chronic heart failure, bleeding disorder, hypertension, chronic renal failure etc.) as determined by their medical history, physical examination, and laboratory studies.
* Body Mass Index (BMI) < 31 kg/m2 (weight/height2).
* Female patients of childbearing potential must have negative pregnancy test within 14 days before initiation of study drug dosing. Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Male and female patients of reproductive potential must agree to employ an effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drug.
* Written, voluntary informed consent.

Exclusion Criteria:

* Abnormal marrow function as defined by leucocyte, neutrophil, or platelet counts outside of normal limits.
* Any evidence of renal dysfunction (proteinuria; serum creatinine > upper limit of normal; or if serum creatinine > upper limit of normal, a calculated creatinine clearance < 60 mL/min/1.73 m2).
* Impaired hepatic function (liver enzymes greater than the upper limit of normal or bilirubin outside the normal range).
* QTcF > 450 msec on screening ECG (using the QTcF formula).
* Patient with electrolyte abnormality (e.g., hypokalemia, hypomagnesemia, hypophosphatemia, hyperkalemia, hypocalcemia, hyponatremia).
* Taking any medications (including over the counter products), herbal products, mineral supplements or vitamins (other than a daily multivitamin preparation), other than contraceptives (for women), within 2 weeks of start of the study. All forms of contraceptive medication are permissible for this study and would not result in a female's exclusion from participation. Patients who take medications on a chronic basis, such as antihypertensive medications or thyroid replacement therapy, etc. are not eligible for the study.
* Subjects has received any other investigational agents within 28 days of first day of study drug dosing.
* Female subjects who are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-11; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To define the effect of administration of a calcium salt (calcium carbonate) on the PK (in particular the area under the nilotinib plasma concentration versus time curve) of nilotinib (Tasigna® ) in healthy volunteers. | PK blood samples are drawn from each subject at time 0 (before each dose of Tasigna®), and at 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, and 72 hrs after adminstration of Tasigna®.

CONTACTS AND LOCATIONS:
Overall Officials: Jan H. Beumer, PharmD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Cancer Institute / Clinical and Translational Research Center (Hillman Cancer Center and Montefiore University Hospital locations), Pittsburgh, Pennsylvania, United States